CLINICAL TRIAL: NCT04492644
Title: The Correlation Among Nutrition, Muscle Strength, Masticatory and Swallow Ability of Inpatient Elders
Acronym: NMM
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yin-Hwa Shih, Assistant professor, China Medical University Hospital
Other Study IDs: CMUH108-REC3-110
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Malnutrition; Moderate
Keywords: the elder inpatient,; nutritional assessment; handgrip strength; masticatory electromyography
MeSH Terms: conditions — Malnutrition; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly inpatients: Elderly inpatients aged 65 years or older who were able to communicate and were clearly conscious. Elderly individuals who were diagnosed with gastrointestinal (GI) dysfunction, dysphagia, edentulism without rehabilitation with dentures, brain disease, stroke or cancer were excluded due to the possibility of dysphagia, cachexia or masticatory muscle palsy.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The masticatory performance would affect the nutritional status of elderly people. the prevalence of undernutrition among elderly inpatients is %20-50%. Previous related studies investigate the masticatory performance with special chewing gum and self-reported questionnaires. This study observes the correlation of masticatory muscles sEMG, nutritional status, and handgrip force among elderly inpatients.

DETAILED DESCRIPTION:
In this cross-sectional study, we enrolled 120 seniors aged 65 and above who are newly admitted to the Asian University Hospital. Within 24 hours they admitted to the hospital, we collected the Mini Nutritional Assessment scores, surface electromyography data, handgrip strength, self-assessment swallowing ability score, and clinical objective data. We performed the statistics for independent t-test, Pearson correlation analysis, and binary logistic regression with SPSS 23 software.

ELIGIBILITY:
Inclusion Criteria:

* new elderly inpatients aged 65 years or older who were able to communicate and were clearly conscious

Exclusion Criteria:

* Elderly individuals who were diagnosed with gastrointestinal (GI) dysfunction, dysphagia, edentulism without rehabilitation with dentures, brain disease, stroke or cancer were excluded due to the possibility of dysphagia, cachexia or masticatory muscle palsy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We enrolled 120 elderly inpatients in Asia University Hospital, Taiwan. We included new elderly inpatients aged 65 years or older who were able to communicate and were clearly conscious.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
masticatory muscle surface EMG | Data were collected after the participants signed the informed consent form within 24 hours admitted to hospital.
  The sEMG examinations were conducted with a Zebris EMG Bluetooth muscle activity recording system

SECONDARY OUTCOMES:
Nutritional status | Data were collected after the participants signed the informed consent form within 24 hours admitted to hospital.
  Nutritional status was measured by the Mini Nutritional Assessment (MNA).

OTHER OUTCOMES:
Handgrip force | Data were collected after the participants signed the informed consent form within 24 hours admitted to hospital.
  Left and right handgrip forces were measured by a Jamar® Hydraulic Hand Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hwa Shih, Ph.D., Principal Investigator — Asia University
Locations (1):
- Asia University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alzahrani SH, Alamri SH. Prevalence of malnutrition and associated factors among hospitalized elderly patients in King Abdulaziz University Hospital, Jeddah, Saudi Arabia. BMC Geriatr. 2017 Jul 3;17(1):136. doi: 10.1186/s12877-017-0527-z. PMID 28673255
- [Result] Berretin-Felix G, Nary Filho H, Padovani CR, Trindade Junior AS, Machado WM. Electromyographic evaluation of mastication and swallowing in elderly individuals with mandibular fixed implant-supported prostheses. J Appl Oral Sci. 2008 Mar-Apr;16(2):116-21. doi: 10.1590/s1678-77572008000200007. PMID 19089202
- [Result] Gomes F, Baumgartner A, Bounoure L, Bally M, Deutz NE, Greenwald JL, Stanga Z, Mueller B, Schuetz P. Association of Nutritional Support With Clinical Outcomes Among Medical Inpatients Who Are Malnourished or at Nutritional Risk: An Updated Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Nov 1;2(11):e1915138. doi: 10.1001/jamanetworkopen.2019.15138. PMID 31747030